CLINICAL TRIAL: NCT00148681
Title: Preoperative Herceptin and Navelbine in Early Stage, HER-2 Positive Breast Cancer
Brief Title: Preoperative Herceptin and Navelbine for Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Eric P Winer, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00-273
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer
Keywords: HER-2 Positive breast cancer; herceptin; navelbine
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Vinorelbine; Doxorubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lower Risk Regimen (Experimental)
  Interventions: Drug: Herceptin; Drug: Navelbine; Drug: Doxorubicin; Drug: Cyclophosphamide
- Higher Risk Regimen (Experimental)
  Interventions: Drug: Herceptin; Drug: Navelbine; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel

INTERVENTIONS:
Drug: Herceptin — Intravenously every week for 12 weeks (weeks 1-12) Intravenously every three weeks for 40 weeks (weeks 32-72)
Drug: Navelbine — Intravenously every week for 12 weeks
Drug: Doxorubicin — Every 3 weeks for 12 weeks
  Other Names: adriamycin
Drug: Cyclophosphamide — Intravenously every 3 weeks for 12 weeks
  Other Names: Cytoxan
Drug: Paclitaxel — Weekly for 12 weeks (or a similar schedule)
  Other Names: Taxol
  Arms: Higher Risk Regimen

SUMMARY:
The purpose of this study is to find out what effects the preoperative combination therapy of herceptin and navelbine have on HER-2 positive breast cancer.

DETAILED DESCRIPTION:
* As part of the patients pre-treatment evaluation, a clip will be placed within the tumor bed so that the surgeon can find it at the time of surgery. Four biopsies of the tumor will be obtained at the time of the clip placement for further testing at a later date.
* Depending upon the patient's risk level (as assessed by the treating physician), they will be treated similarly to one of two regimens. The first 8 months of both regimens are the same consisting of 12 weeks of herceptin and navelbine, followed by surgery and then 4 cycles of adriamycin and cytoxan. The treatment following these 8 months will depend upon the health risk to the patient and will be determined by both the patient and treating physician.
* Group 1: Lower Risk Regimen: Patients in this group will receive 3 phases of treatment. In Phase A they will receive Navelbine and Herceptin intravenously every week for 12 weeks. Upon completion of this therapy they will undergo surgery to remove the tumor. Following surgery there will be a 6 week recovery period where no treatment will be received. In Phase B, patients will receive adriamycin (doxorubicin) and cytoxan (cyclophosphamide) intravenously every 3 weeks for 12 weeks, for a total of 4 cycles. Patients then may or may not receive Phase C (depending upon physicians discretion), during which they will receive herceptin intravenously every 3 weeks for 40 weeks. If the physician decides that the patient needs radiation therapy, it will commence after the completion of adriamycin and cytoxan.
* Group 2: Higher Risk Regimen: Patients in this group will undergo four different phases of treatment. Phase A is identical to that of Group 1 (herceptin and navelbine for 12 weeks followed by surgery) as is Phase B (adriamycin and cytoxan every 3 weeks for 12 weeks for a total of 4 cycles). Phase C will consist of paclitaxel and herceptin weekly for a total of 12 weeks. If the physician decides that radiation therapy should be performed, it will commence within 6 weeks of the last dose of paclitaxel and herceptin. In Phase D, patients will receive herceptin intravenously every three weeks for 28 weeks.
* The following procedures and tests will be performed during this study: During Phase A: Every week: blood work; Every 3 weeks: physical exam, tumor assessment and bloodwork. During Phase B: Every 3 weeks; physical exam and blood work. At the start of Phase B and C: physical exam, EKG, MUGA scan or echocardiogram and bloodwork. During Phase C: Every 3 weeks for High risk patients and every 3 months for low risk patients; physical exam and blood work. End of Phase C: MUGA scan or echocardiogram. Phase C and D: every 3 months; physical exam, EGK, MUGA scan or echocardiogram and bloodwork.
* At the end of the study patients will undergo a physical exam, EKG, MUGA scan or echocardiogram and bloodwork.

ELIGIBILITY:
Inclusion Criteria:

* EGOG performance status of 0-1
* HER2 overexpressing (IHC 3+ or FISH +)
* Stage II or III breast cancer. Clinical T1N1M) and inflammatory (T4) breast cancer are eligible
* Patients with metastatic breast cancer (Stage IV) which is limited to supraclavicular and/or infraclavicular node positivity are eligible
* 18 years of age or older

Exclusion Criteria:

* Prior therapy with herceptin, paclitaxel or other taxane, doxorubicin or other anthracycline-type chemotherapy, navelbine
* Pregnant or lactating women
* Uncontrolled infections, including AIDS
* History or symptoms diagnostic of systemic connective tissue or inflammatory disease
* Active or severe cardiovascular or pulmonary disease, including recent myocardial infarction or deep-venous thrombosis/pulmonary embolism, congestive heart failure, uncontrolled hypertension, or steroid-dependent asthma.
* Left ventricular ejection fraction < 50%
* Peripheral neuropathy of any etiology that exceeds grade 1
* Prior history of malignancy treated without curative intent
* Uncontrolled diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2001-05; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
To assess the complete response rate after preoperative herceptin and navelbine in HER-2 positive breast cancer. | 2 years

SECONDARY OUTCOMES:
To determine the safety of herceptin and navelbine in this patient population (either high risk or low risk). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Winer, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Center, Boston, Massachusetts